CLINICAL TRIAL: NCT05284760
Title: A Phase 1, Open-Label, Randomized, Crossover Study to Evaluate the Bioequivalence of Soticlestat Oral Tablet Formulations and the Effect of Food and Tablet Crushing on the Pharmacokinetics of Soticlestat in Healthy Adult Participants
Brief Title: A Study of Soticlestat Tablets in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: TAK-935-1014
Record Dates: First submitted 2022-03-10; First posted 2022-03-17 (Actual); Results first posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy
MeSH Terms: interventions — soticlestat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (12):
- Part A, Sequence 1: Treatment A + Treatment B + Treatment C (Experimental): Soticlestat T4 tablets 300 mg, orally, once on Day 1 of Period 1 under fasted condition as Treatment A, followed by soticlestat T3 mini-tablets 300 mg, orally, once on Day 1 of Period 2 under fasted condition as Treatment B, and followed by soticlestat T3 commercial tablets 300 mg, orally, once on Day 1 of Period 3 under fasted condition as Treatment C. A washout interval of exactly 4 days will be maintained between each Treatment Period.
  Interventions: Drug: Soticlestat
- Part A, Sequence 2: Treatment A + Treatment C + Treatment B (Experimental): Soticlestat T4 tablets 300 mg, orally, once on Day 1 of Period 1 under fasted condition as Treatment A, followed by soticlestat T3 commercial tablets 300 mg, orally, once on Day 1 of Period 2 under fasted condition as Treatment C, and followed by soticlestat T3 mini-tablets 300 mg, orally, once on Day 1 of Period 3 under fasted condition as Treatment B. A washout interval of exactly 4 days will be maintained between each Treatment Period.
  Interventions: Drug: Soticlestat
- Part A, Sequence 3: Treatment B + Treatment A + Treatment C (Experimental): Soticlestat T3 mini-tablets 300 milligram (mg), orally, once on Day 1 of Period 1 under fasted condition as Treatment B, followed by soticlestat T4 300 mg, tablets, orally, once on Day 1 of Period 2 under fasted condition as Treatment A, and followed by soticlestat T3 commercial tablets 300 mg, orally, once on Day 1 of Period 3 under fasted condition as Treatment C. A washout interval of exactly 4 days will be maintained between each Treatment Period.
  Interventions: Drug: Soticlestat
- Part A, Sequence 4: Treatment B + Treatment C + Treatment A (Experimental): Soticlestat T3 mini-tablets 300 mg, orally, once on Day 1 of Period 1 under fasted condition as Treatment B, followed by soticlestat T3 commercial tablets 300 mg, orally, once on Day 1 of Period 2 under fasted condition as Treatment C, and followed by soticlestat T4 300 mg, tablets, orally, once on Day 1 of Period 3 under fasted condition as Treatment A. A washout interval of exactly 4 days will be maintained between each Treatment Period.
  Interventions: Drug: Soticlestat
- Part A, Sequence 5: Treatment C + Treatment A + Treatment B (Experimental): Soticlestat T3 commercial tablets 300 mg, orally, once on Day 1 of Period 1 under fasted condition as Treatment C, followed by soticlestat T4 300 mg, tablets, orally, once on Day 1 of Period 2 under fasted condition as Treatment A, and followed by soticlestat T3 mini-tablets 300 mg, orally, once on Day 1 of Period 3 under fasted condition as Treatment B. A washout interval of exactly 4 days will be maintained between each Treatment Period.
  Interventions: Drug: Soticlestat
- Part A, Sequence 6: Treatment C + Treatment B + Treatment A (Experimental): Soticlestat T3 commercial tablets 300 mg, orally, once on Day 1 of Period 1 under fasted condition as Treatment C, followed by soticlestat T3 mini-tablets 300 mg, tablets, orally, once on Day 1 of Period 2 under fasted condition as Treatment B, and followed by soticlestat T4 tablets 300 mg, orally, once on Day 1 of Period 3 under fasted condition as Treatment A. A washout interval of exactly 4 days will be maintained between each Treatment Period.
  Interventions: Drug: Soticlestat
- Part B, Sequence 1: Treatment D + Treatment E + Treatment F (Experimental): Soticlestat T4 300 mg, tablets, orally, once on Day 1 of Period 1 under fasted condition as Treatment D, followed by soticlestat T4 300 mg, tablets, orally, once on Day 1 of Period 2 under fed condition as Treatment E, and followed by soticlestat T4 300 mg tablets crushed and mixed with applesauce, orally, once on Day 1 of Period 3 under fasted condition as Treatment F. A washout interval of exactly 4 days will be maintained between each Treatment Period.
  Interventions: Drug: Soticlestat
- Part B, Sequence 2: Treatment D + Treatment F + Treatment E (Experimental): Soticlestat T4 300 mg, tablets, orally, once on Day 1 of Period 1 under fasted condition as Treatment D, followed by soticlestat T4 300 mg, tablets crushed and mixed with applesauce, orally, once on Day 1 of Period 2 under fasted condition as Treatment F, and followed by soticlestat T4 300 mg, orally, once on Day 1 of Period 3 under fed condition as Treatment E. A washout interval of exactly 4 days will be maintained between each Treatment Period.
  Interventions: Drug: Soticlestat
- Part B, Sequence 3: Treatment E + Treatment D + Treatment F (Experimental): Soticlestat T4 300 mg, tablets, orally, once on Day 1 of Period 1 under fed condition as Treatment E, followed by soticlestat T4 300 mg, tablets, orally, once on Day 1 of Period 2 under fasted condition as Treatment D, and followed by soticlestat T4 300 mg, tablets crushed and mixed with applesauce, orally, once on Day 1 of Period 3 under fasted condition as Treatment F. A washout interval of exactly 4 days will be maintained between each Treatment Period.
  Interventions: Drug: Soticlestat
- Part B, Sequence 4: Treatment E + Treatment F + Treatment D (Experimental): Soticlestat T4 300 mg, tablets, orally, once on Day 1 of Period 1 under fed condition as Treatment E, followed by soticlestat T4 300 mg tablets crushed and mixed with applesauce, orally, once on Day 1 of Period 2 under fasted condition as Treatment F, and followed by soticlestat T4 300 mg, tablets, orally, once on Day 1 of Period 3 under fasted condition as Treatment D. A washout interval of exactly 4 days will be maintained between each Treatment Period.
  Interventions: Drug: Soticlestat
- Part B, Sequence 5: Treatment F + Treatment D + Treatment E (Experimental): Soticlestat T4 300 mg tablets crushed and mixed with applesauce, orally, once on Day 1 of Period 1 under fasted condition as Treatment F, followed by soticlestat T4 300 mg, tablets, orally, once on Day 1 of Period 2 under fasted condition as Treatment D, and followed by soticlestat T4 300 mg, tablets, orally, once on Day 1 of Period 3 under fed condition as Treatment E. A washout interval of exactly 4 days will be maintained between each Treatment Period.
  Interventions: Drug: Soticlestat
- Part B, Sequence 3: Treatment F + Treatment E + Treatment D (Experimental): Soticlestat T4 300 mg tablets, crushed and mixed with applesauce, orally, once on Day 1 of Period 1 under fasted condition as Treatment F, followed by soticlestat T4 300 mg, tablets, orally, once on Day 1 of Period 2 under fed condition as Treatment E, and followed by soticlestat T4 300 mg tablets, orally, once on Day 1 of Period 3 under fasted condition as Treatment D. A washout interval of exactly 4 days will be maintained between each Treatment Period.
  Interventions: Drug: Soticlestat

INTERVENTIONS:
Drug: Soticlestat — Soticlestat T4 tablets.
  Other Names: TAK-935
Drug: Soticlestat — Soticlestat T3 mini-tablets.
  Other Names: TAK-935
Drug: Soticlestat — Soticlestat commercial tablets.
  Other Names: TAK-935

SUMMARY:
The main aim is to see how soticlestat tablets of different strengths work and to compare how it works alone in contrast to administration along with food.

In the study will be 2 groups of participants (part A and part B). Participants in part A will receive 300 mg of soticlestat administered in different kind of tablets (regular tablets, mini-tablets, commercial tablets) and participant in part B will also receive 300 mg of soticlestat in tablets but with food and crushed tablets with applesauce.

Participants will complete several assessments including clinical laboratory evaluations, physical examinations, Columbia-Suicide Severity Rating Scale (C-SSRS) assessment, electrocardiographs (ECGs), and vital signs.

DETAILED DESCRIPTION:
The drug being tested in this study is called soticlestat (TAK-935). The study will assess the bioequivalence, effect of food and tablet crushing, safety and tolerability following single oral dose of 3 different soticlestat oral tablet formulations in healthy participants.

The study will enroll approximately 96 participants. This study will be conducted in two parts (Part A and Part B) having 6 treatment sequences each. Participants will be randomly assigned (by chance, like flipping a coin) to one of the study parts as per treatment sequence:

* Part A, Sequence 1: Treatment A + Treatment B + Treatment C
* Part A, Sequence 2: Treatment A + Treatment C + Treatment B
* Part A, Sequence 3: Treatment B + Treatment A + Treatment C
* Part A, Sequence 4: Treatment B + Treatment C + Treatment A
* Part A, Sequence 5: Treatment C + Treatment A + Treatment B
* Part A, Sequence 6: Treatment C + Treatment B + Treatment A
* Part B, Sequence 1: Treatment D + Treatment E + Treatment F
* Part B, Sequence 2: Treatment D + Treatment F + Treatment E
* Part B, Sequence 3: Treatment E + Treatment D + Treatment F
* Part B, Sequence 4: Treatment E + Treatment F + Treatment D
* Part B, Sequence 5: Treatment F + Treatment D + Treatment E
* Part B, Sequence 6: Treatment F + Treatment E + Treatment D

This single center trial will be conducted in the United States. The overall duration of the study is approximately 51 days. Participants will be followed up for 14 days after the last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Key Inclusion Criteria:

1. Body mass index (BMI) greater than or equal to (>=) 18.0 and less than or equal to (<=) 32.0 kilogram per square meter (kg/m^2) at screening.
2. Continuous non-smoker who has not used nicotine-containing products for at least 90 days prior to the first dosing.
3. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs, and ECGs, as deemed by the Investigator or designee.
4. Able to swallow multiple tablets.

Key Exclusion Criteria:

1. History or presence of alcoholism or drug abuse within the past 2 years prior to the first dosing.
2. Positive urine drug or alcohol results at screening or check-in.
3. Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV).
4. Unable to refrain from or anticipates the use of:

   * Any drug, including prescription and non-prescription medications, herbal remedies, or vitamin supplements within 14 days prior to the first dosing. Thyroid hormone replacement medication may be permitted if the participant has been on the same stable dose for the immediate 3 months prior to the first dosing.
   * Any drugs known to be significant inducers of cytochrome P450 (CYP) 3A, CYP2C19, uridine 5'-diphospho-glucuronosyltransferase (UGT) 1A9 or UGT2B4 enzymes and/or P-glycoprotein (P-gp), including St. John's Wort, within 28 days prior to the first dosing. Appropriate sources will be consulted to confirm lack of PK/pharmacodynamics interaction with study drug.
5. History of alcohol consumption exceeding 2 standard drinks per day on average (1 glass is approximately equivalent to the following: beer [354 milliliter per 12 ounce {mL/12 oz}], wine [118 mL/4 oz], or distilled spirits [29.5 mL/1 oz] per day).
6. Consumes excessive amounts, defined as greater than 4 servings (1 serving is approximately equivalent to 120mg of caffeine), of coffee, tea, cola, energy drinks, or other caffeinated beverages per day.
7. Has been on a diet incompatible with the on-study diet, in the opinion of the Investigator or designee, within the 30 days prior to the first dosing and throughout the study.
8. Donation of blood or significant blood loss within 56 days prior to the first dosing.
9. Plasma donation within 7 days prior to the first dosing.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2022-05-22 (Actual); Study Completion 2022-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/30b7d725c12c42a5?idFilter=%5B%22TAK-935-1014%22%5D

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A, Sequence 1: Treatment A + Treatment B + Treatment C: Soticlestat T4 tablets 300 mg, orally, once on Day 1 of Period 1 under fasted condition as Treatment A, followed by soticlestat T3 mini-tablets 300 mg, orally, once on Day 1 of Period 2 under fasted condition as Treatment B, and followed by soticlestat T3 commercial tablets 300 mg, orally, once on Day 1 of Period 3 under fasted condition as Treatment C. A washout interval of exactly 4 days was maintained between each Treatment Period.
- Part A, Sequence 2: Treatment A + Treatment C + Treatment B: Soticlestat T4 tablets 300 mg, orally, once on Day 1 of Period 1 under fasted condition as Treatment A, followed by soticlestat T3 commercial tablets 300 mg, orally, once on Day 1 of Period 2 under fasted condition as Treatment C, and followed by soticlestat T3 mini-tablets 300 mg, orally, once on Day 1 of Period 3 under fasted condition as Treatment B. A washout interval of exactly 4 days was maintained between each Treatment Period.
- Part A, Sequence 3: Treatment B + Treatment A + Treatment C: Soticlestat T3 mini-tablets 300 milligram (mg), orally, once on Day 1 of Period 1 under fasted condition as Treatment B, followed by soticlestat T4 300 mg, tablets, orally, once on Day 1 of Period 2 under fasted condition as Treatment A, and followed by soticlestat T3 commercial tablets 300 mg, orally, once on Day 1 of Period 3 under fasted condition as Treatment C. A washout interval of exactly 4 days was maintained between each Treatment Period.
- Part A, Sequence 4: Treatment B + Treatment C + Treatment A: Soticlestat T3 mini-tablets 300 mg, orally, once on Day 1 of Period 1 under fasted condition as Treatment B, followed by soticlestat T3 commercial tablets 300 mg, orally, once on Day 1 of Period 2 under fasted condition as Treatment C, and followed by soticlestat T4 300 mg, tablets, orally, once on Day 1 of Period 3 under fasted condition as Treatment A. A washout interval of exactly 4 days was maintained between each Treatment Period.
- Part A, Sequence 5: Treatment C + Treatment A + Treatment B: Soticlestat T3 commercial tablets 300 mg, orally, once on Day 1 of Period 1 under fasted condition as Treatment C, followed by soticlestat T4 300 mg, tablets, orally, once on Day 1 of Period 2 under fasted condition as Treatment A, and followed by soticlestat T3 mini-tablets 300 mg, orally, once on Day 1 of Period 3 under fasted condition as Treatment B. A washout interval of exactly 4 days was maintained between each Treatment Period.
- Part A, Sequence 6: Treatment C + Treatment B + Treatment A: Soticlestat T3 commercial tablets 300 mg, orally, once on Day 1 of Period 1 under fasted condition as Treatment C, followed by soticlestat T3 mini-tablets 300 mg, tablets, orally, once on Day 1 of Period 2 under fasted condition as Treatment B, and followed by soticlestat T4 tablets 300 mg, orally, once on Day 1 of Period 3 under fasted condition as Treatment A. A washout interval of exactly 4 days was maintained between each Treatment Period.
- Part B, Sequence 1: Treatment D + Treatment E + Treatment F: Soticlestat T4 300 mg, tablets, orally, once on Day 1 of Period 1 under fasted condition as Treatment D, followed by soticlestat T4 300 mg, tablets, orally, once on Day 1 of Period 2 under fed condition as Treatment E, and followed by soticlestat T4 300 mg tablets crushed and mixed with applesauce, orally, once on Day 1 of Period 3 under fasted condition as Treatment F. A washout interval of exactly 4 days was maintained between each Treatment Period.
- Part B, Sequence 2: Treatment D + Treatment F + Treatment E: Soticlestat T4 300 mg, tablets, orally, once on Day 1 of Period 1 under fasted condition as Treatment D, followed by soticlestat T4 300 mg, tablets crushed and mixed with applesauce, orally, once on Day 1 of Period 2 under fasted condition as Treatment F, and followed by soticlestat T4 300 mg, orally, once on Day 1 of Period 3 under fed condition as Treatment E. A washout interval of exactly 4 days was maintained between each Treatment Period.
- Part B, Sequence 3: Treatment E + Treatment D + Treatment F: Soticlestat T4 300 mg, tablets, orally, once on Day 1 of Period 1 under fed condition as Treatment E, followed by soticlestat T4 300 mg, tablets, orally, once on Day 1 of Period 2 under fasted condition as Treatment D, and followed by soticlestat T4 300 mg, tablets crushed and mixed with applesauce, orally, once on Day 1 of Period 3 under fasted condition as Treatment F. A washout interval of exactly 4 days was maintained between each Treatment Period.
- Part B, Sequence 4: Treatment E + Treatment F + Treatment D: Soticlestat T4 300 mg, tablets, orally, once on Day 1 of Period 1 under fed condition as Treatment E, followed by soticlestat T4 300 mg tablets crushed and mixed with applesauce, orally, once on Day 1 of Period 2 under fasted condition as Treatment F, and followed by soticlestat T4 300 mg, tablets, orally, once on Day 1 of Period 3 under fasted condition as Treatment D. A washout interval of exactly 4 days was maintained between each Treatment Period.
- Part B, Sequence 5: Treatment F + Treatment D + Treatment E: Soticlestat T4 300 mg tablets crushed and mixed with applesauce, orally, once on Day 1 of Period 1 under fasted condition as Treatment F, followed by soticlestat T4 300 mg, tablets, orally, once on Day 1 of Period 2 under fasted condition as Treatment D, and followed by soticlestat T4 300 mg, tablets, orally, once on Day 1 of Period 3 under fed condition as Treatment E. A washout interval of exactly 4 days was maintained between each Treatment Period.
- Part B, Sequence 6: Treatment F + Treatment E + Treatment D: Soticlestat T4 300 mg tablets, crushed and mixed with applesauce, orally, once on Day 1 of Period 1 under fasted condition as Treatment F, followed by soticlestat T4 300 mg, tablets, orally, once on Day 1 of Period 2 under fed condition as Treatment E, and followed by soticlestat T4 300 mg tablets, orally, once on Day 1 of Period 3 under fasted condition as Treatment D. A washout interval of exactly 4 days was maintained between each Treatment Period.
Period: Overall Study
Arm/Group | Part A, Sequence 1: Treatment A + Treatment B + Treatment C | Part A, Sequence 2: Treatment A + Treatment C + Treatment B | Part A, Sequence 3: Treatment B + Treatment A + Treatment C | Part A, Sequence 4: Treatment B + Treatment C + Treatment A | Part A, Sequence 5: Treatment C + Treatment A + Treatment B | Part A, Sequence 6: Treatment C + Treatment B + Treatment A | Part B, Sequence 1: Treatment D + Treatment E + Treatment F | Part B, Sequence 2: Treatment D + Treatment F + Treatment E | Part B, Sequence 3: Treatment E + Treatment D + Treatment F | Part B, Sequence 4: Treatment E + Treatment F + Treatment D | Part B, Sequence 5: Treatment F + Treatment D + Treatment E | Part B, Sequence 6: Treatment F + Treatment E + Treatment D
Started | 12 | 12 | 12 | 12 | 12 | 12 | 4 | 4 | 4 | 4 | 4 | 4
Completed | 12 | 12 | 12 | 12 | 12 | 12 | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of the study drug(s) were included in the safety set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A, Sequence 1: Treatment A + Treatment B + Treatment C | Part A, Sequence 2: Treatment A + Treatment C + Treatment B | Part A, Sequence 3: Treatment B + Treatment A + Treatment C | Part A, Sequence 4: Treatment B + Treatment C + Treatment A | Part A, Sequence 5: Treatment C + Treatment A + Treatment B | Part A, Sequence 6: Treatment C + Treatment B + Treatment A | Part B, Sequence 1: Treatment D + Treatment E + Treatment F | Part B, Sequence 2: Treatment D + Treatment F + Treatment E | Part B, Sequence 3: Treatment E + Treatment D + Treatment F | Part B, Sequence 4: Treatment E + Treatment F + Treatment D | Part B, Sequence 5: Treatment F + Treatment D + Treatment E | Part B, Sequence 6: Treatment F + Treatment E + Treatment D | Total
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 4 | 4 | 4 | 4 | 4 | 4 | 96
Age, Continuous [Mean (Full Range); unit: years] | 41.1 [29 to 54] | 38.3 [26 to 52] | 43.1 [20 to 55] | 38.3 [22 to 54] | 40.4 [25 to 54] | 40.3 [28 to 53] | 40.0 [36 to 52] | 37.8 [32 to 44] | 49.5 [46 to 53] | 42.3 [35 to 49] | 30.3 [20 to 50] | 38.3 [30 to 45] | 40.1 [20 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 1 | 5 | 3 | 3 | 1 | 1 | 0 | 1 | 0 | 1 | 23
  Male | 8 | 9 | 11 | 7 | 9 | 9 | 3 | 3 | 4 | 3 | 4 | 3 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 8 | 7 | 10 | 10 | 9 | 4 | 4 | 4 | 4 | 4 | 2 | 75
  Not Hispanic or Latino | 3 | 4 | 5 | 2 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 2 | 21
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 3 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 10
  White | 12 | 9 | 9 | 11 | 10 | 12 | 4 | 3 | 4 | 3 | 4 | 4 | 85
  More than one race | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Full Range); unit: kilogram per meters squared (kg/m^2)] — BMI was calculated based on the height and weight, using the formula: BMI = weight (kg)/[height (m)^2].
  kilogram per meters squared (kg/m^2) | 26.626 [21.23 to 31.28] | 27.249 [22.97 to 31.23] | 27.859 [25.48 to 30.85] | 27.943 [24.07 to 31.68] | 26.840 [20.89 to 30.97] | 26.626 [21.23 to 31.28] | 26.843 [24.61 to 28.18] | 26.285 [23.49 to 29.24] | 28.030 [25.76 to 31.62] | 27.120 [24.98 to 29.10] | 26.130 [22.07 to 28.27] | 26.960 [23.58 to 30.91] | 27.286 [20.89 to 31.68]
Height [Mean (Full Range); unit: centimeters (cm)] | 166.8 [153 to 189] | 169.4 [154 to 179] | 174.8 [161 to 185] | 167.5 [151 to 191] | 171.8 [156 to 186] | 168.5 [151 to 184] | 172.3 [167 to 175] | 171.8 [159 to 182] | 172.0 [171 to 173] | 168.0 [155 to 180] | 172.0 [167 to 177] | 170.0 [158 to 181] | 170.1 [151 to 191]
Weight [Mean (Full Range); unit: kg] | 74.09 [58.1 to 98.7] | 78.38 [54.4 to 95.7] | 85.33 [68.4 to 100.4] | 78.12 [64.1 to 92.9] | 78.83 [63.4 to 97.0] | 79.67 [60.4 to 98.2] | 79.35 [75.4 to 82.5] | 77.33 [68.1 to 87.5] | 82.90 [76.4 to 92.4] | 77.03 [63.7 to 90.1] | 77.78 [61.8 to 88.9] | 78.80 [62.6 to 101.4] | 79.02 [54.4 to 101.4]

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for Soticlestat
Time Frame: Day 1 pre-dose and at multiple time points (up to 96 hours) post-dose
Population: All participants who complied sufficiently with the protocol and displayed an evaluable Pharmacokinetic (PK) profile (eg, exposure to treatment, availability of measurements, and absence of major protocol violations) were included in the PK set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milllilitre (ng/ml)
Groups:
- Part A - Treatment A: Soticlestat T4 tablets 300 mg, orally, once on Day 1 of each period under fasted condition.
- Part A - Treatment B: Soticlestat T3 mini-tablets 300 mg, orally, once on Day 1 of each period under fasted condition.
- Part A - Treatment C: Soticlestat T3 commercial tablets 300 mg, orally, once on Day 1 of each period under fasted condition.
- Part B - Treatment D: Soticlestat T4 300 mg, tablets, orally, once on Day 1 of each period under fasted condition.
- Part B - Treatment E: Soticlestat T4 300 mg, tablets, orally, once on Day 1 of each period under fed condition.
- Part B - Treatment F: Soticlestat T4 300 mg, tablets crushed and mixed with applesauce, orally, once on Day 1 of each period under fasted condition.
Arm/Group | Part A - Treatment A | Part A - Treatment B | Part A - Treatment C | Part B - Treatment D | Part B - Treatment E | Part B - Treatment F
Number analyzed (Participants) | 72 | 72 | 71 | 24 | 24 | 24
nanogram per milllilitre (ng/ml) | 1762 (66.3) | 1428 (76.0) | 1708 (65.1) | 1509 (65.7) | 565.6 (49.0) | 1350 (63.1)
Statistical Analysis 1: Comparison: Part A - Treatment A vs Part A - Treatment C; Test type: Equivalence — The two treatments were deemed equivalent if the 90% CIs for the GMRs for all of the parameters were each within 80.00% and 125.00%; Geometric Mean Ratio (GMR) = 97.28, 90% CI 2-sided [87.66 to 107.96]
Statistical Analysis 2: Comparison: Part A - Treatment A vs Part A - Treatment B; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; GMR = 81.04, 90% CI 2-sided [73.06 to 89.89]
Statistical Analysis 3: Comparison: Part B - Treatment D vs Part B - Treatment E; Test type: Other; GMR = 37.48, 90% CI 2-sided [31.10 to 45.17]
Statistical Analysis 4: Comparison: Part B - Treatment D vs Part B - Treatment F; Test type: Other; GMR = 89.45, 90% CI 2-sided [74.24 to 107.79]

2. Primary Outcome: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Soticlestat
Time Frame: Day 1 pre-dose and at multiple time points (up to 96 hours) post-dose
Population: All participants who complied sufficiently with the protocol and displayed an evaluable PK profile (eg, exposure to treatment, availability of measurements, and absence of major protocol violations) were included in the PK set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.hour (hr)/ml
Arm/Group | Part A - Treatment A | Part A - Treatment B | Part A - Treatment C | Part B - Treatment D | Part B - Treatment E | Part B - Treatment F
Number analyzed (Participants) | 72 | 72 | 71 | 24 | 24 | 24
ng.hour (hr)/ml | 1649 (50.2) | 1433 (54.8) | 1606 (51.6) | 1503 (49.1) | 1317 (37.0) | 1435 (61.9)
Statistical Analysis 1: Comparison: Part A - Treatment A vs Part A - Treatment C; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; GMR = 97.52, 90% CI 2-sided [92.17 to 103.17]
Statistical Analysis 2: Comparison: Part A - Treatment A vs Part A - Treatment B; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; GMR = 86.88, 90% CI 2-sided [82.14 to 91.89]
Statistical Analysis 3: Comparison: Part B - Treatment D vs Part B - Treatment E; Test type: Other; GMR = 87.63, 90% CI 2-sided [75.92 to 101.15]
Statistical Analysis 4: Comparison: Part B - Treatment D vs Part B - Treatment F; Test type: Other; GMR = 95.49, 90% CI 2-sided [82.73 to 110.22]

3. Primary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for Soticlestat
Time Frame: Day 1 pre-dose and at multiple time points (up to 96 hours) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.hr/ml
Arm/Group | Part A - Treatment A | Part A - Treatment B | Part A - Treatment C | Part B - Treatment D | Part B - Treatment E | Part B - Treatment F
Number analyzed (Participants) | 62 | 55 | 56 | 22 | 22 | 21
ng.hr/ml | 1659 (51.0) | 1459 (58.1) | 1639 (53.7) | 1525 (50.6) | 1354 (35.1) | 1395 (49.6)
Statistical Analysis 1: Comparison: Part A - Treatment A vs Part A - Treatment C; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; GMR = 99.25, 90% CI 2-sided [92.84 to 106.10]
Statistical Analysis 2: Comparison: Part A - Treatment A vs Part A - Treatment B; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; GMR = 86.98, 90% CI 2-sided [81.33 to 93.03]
Statistical Analysis 3: Comparison: Part B - Treatment D vs Part B - Treatment E; Test type: Other; GMR = 89.28, 90% CI 2-sided [78.92 to 100.99]
Statistical Analysis 4: Comparison: Part B - Treatment D vs Part B - Treatment F; Test type: Other; GMR = 92.77, 90% CI 2-sided [81.77 to 105.25]

4. Secondary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: From screening up to 14 days after the last dose of soticlestat (Day 51)
Population: All participants who received at least one dose of the study drug(s) were included in the safety set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - Treatment A | Part A - Treatment B | Part A - Treatment C | Part B - Treatment D | Part B - Treatment E | Part B - Treatment F
Number analyzed (Participants) | 72 | 72 | 72 | 24 | 24 | 24
Participants | 6 | 12 | 7 | 0 | 2 | 1

ADVERSE EVENTS:
Time Frame: From screening up to 14 days after the last dose of soticlestat (Day 51)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Groups:
- Part A: Treatment A: Soticlestat T4 tablets 300 mg, orally, once on Day 1 of each period under fasted condition.
- Part A: Treatment B: Soticlestat T3 mini-tablets 300 mg, orally, once on Day 1 of each period under fasted condition.
- Part A: Treatment C: Soticlestat T3 commercial tablets 300 mg, orally, once on Day 1 of each period under fasted condition.
- Part B: Treatment D: Soticlestat T4 300 mg, tablets, orally, once on Day 1 of each period under fasted condition.
- Part B: Treatment E: Soticlestat T4 300 mg, tablets, orally, once on Day 1 of each period under fed condition.
- Part B: Treatment F: Soticlestat T4 300 mg, tablets crushed and mixed with applesauce, orally, once on Day 1 of each period under fasted condition.
Arm/Group | Part A: Treatment A | Part A: Treatment B | Part A: Treatment C | Part B: Treatment D | Part B: Treatment E | Part B: Treatment F
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/72 | 0/72 | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/72 | 0/72 | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 4/72 | 5/72 | 0/72 | 0/24 | 2/24 | 1/24
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Treatment A (N=72) | Part A: Treatment B (N=72) | Part A: Treatment C (N=72) | Part B: Treatment D (N=24) | Part B: Treatment E (N=24) | Part B: Treatment F (N=24)
Constipation (Gastrointestinal disorders) | 3 | 2 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 3 | 0 | 0 | 1 | 1
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results was made without Sponsor's prior written approval. Any proposed publication or presentation was submitted to Sponsor for review 60 days in advance of publication. Institution will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for an additional 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/60/NCT05284760/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-22): https://cdn.clinicaltrials.gov/large-docs/60/NCT05284760/SAP_001.pdf